CLINICAL TRIAL: NCT06043778
Title: Digital Implementation Support to Achieve Uptake and Integration of Task-Shared Care for Schizophrenia in Primary Care in India
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Sangath (Other); National Institute of Mental Health and Neuro Sciences, India (Other); All India Institute of Medical Sciences, Bhopal (Other)
Responsible Party: Principal Investigator, John A. Naslund, Instructor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH133230 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Schizophrenia and Related Disorders; Psychosocial Functioning
Keywords: schizophrenia; psychosocial intervention; digital technology; task sharing; implementation; smartphone app
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this trial, the Outcome Assessors administering study assessments at baseline, midpoints and the endpoint will be masked to the intervention arm that participants are allocated to receive. The Study Investigators will also be masked to the intervention arm that participants are allocated to receive. Masking Outcome Assessors and Study Investigators will minimize potential bias due to knowledge of which arm the participant is allocated to, and can ensure unbiased ascertainment of study outcomes is possible. For allocation concealment, the intervention allocation for each participant will not be revealed to the participant until they have been enrolled into the trial, to avoid selection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPSI plus mindLAMP (Experimental): Participants allocated to this arm will be enrolled in COPSI and also have access to the mindLAMP mobile application. mindLAMP's materials will be available on demand for participants use.
  Interventions: Behavioral: Community care for People with Schizophrenia in India (COPSI); Behavioral: mindLAMP Mobile Application
- COPSI (Active Comparator): Participants allocated to this arm will be enrolled in COPSI alone. COPSI is delivered in three phases: 1) intensive engagement (0-3 months), including six to eight home visits by Community Health Officers; 2) stabilization phase (4-7 months) with sessions delivered once every 15 days; 3) and maintenance phase (8-12) with sessions delivered once a month.
  Interventions: Behavioral: Community care for People with Schizophrenia in India (COPSI)

INTERVENTIONS:
Behavioral: Community care for People with Schizophrenia in India (COPSI) — This intervention is designed to promote collaboration between the person with schizophrenia, their caregivers and the treatment team to deliver a flexible, individualized, and needs-based intervention. The COPSI intervention will be delivered by Community Health Officers in three phases: intensive engagement (0-3 months), stabilization phase (4-7 months), and maintenance phase (8-12).
  Other Names: Psychosocial rehabilitation intervention
Behavioral: mindLAMP Mobile Application — Participants in COPSI plus mindLAMP arm will have access to COPSI and the mindLAMP mobile application. mindLAMP has already been co-developed and culturally adapted by patients, family members, and clinicians at both Indian sites. Materials (articles, videos, web links, audio files, etc.) will be available on-demand and can be accessed by patients at any time. Community Health Officers will also schedule content to specific participants to promote engagement.
  Arms: COPSI plus mindLAMP

SUMMARY:
Schizophrenia represents a significant contributor to the global burden of disease, with this burden disproportionately impacting low- and middle-income countries (LMICs). In India, the burden due to schizophrenia is further exacerbated by low access to effective psychosocial interventions aimed at promoting recovery, rehabilitation, and community tenure, as well as inadequate attention to managing co-occurring chronic medical conditions that result in significantly reduced life expectancy among those living with schizophrenia compared to the general population. A major driver of these alarming gaps in access to care for persons with schizophrenia in India is the limited capacity within primary care settings aimed at addressing the complex co-occurring mental health, physical health, and functional needs of this patient population. There now exists strong evidence demonstrating that community programs delivered in primary care and leveraging psychosocial interventions combined with linkage to specialty psychiatric services are effective for supporting treatment and recovery of schizophrenia in low-resource settings. We will leverage our existing collaboration and robust research infrastructure in both rural and urban settings in Madhya Pradesh and Karnataka, India to conduct a hybrid type 1 effectiveness-implementation trial to evaluate whether the use of a digital platform offers added clinical benefit and can support integration of this task shared care for schizophrenia into routine primary care settings. We will address the following aims: 1) evaluate whether the use of the mindLAMP digital platform can enhance the clinical effectiveness of task-shared community-based psychosocial rehabilitation (COPSI) for individuals with schizophrenia, and 2) determine whether the addition of mindLAMP to the delivery of the COPSI program has an impact on implementation metrics when compared to delivery of COPSI alone.

DETAILED DESCRIPTION:
Schizophrenia is one of the leading causes of disability due to mental disorders in low-income and middle-income countries (LMICs), such as India, with this burden disproportionately impacting lower income individuals who primarily access health care services through publicly run facilities. In 2017, it was estimated that there were over 3.5 million people in India living with schizophrenia, with an increasing prevalence of schizophrenia observed from 1990 to 2017 as the population ages and disease burden shifts to chronic conditions experienced in adulthood. Importantly, the burden of disability due to schizophrenia is often underestimated as many epidemiological studies do not adequately account for the added burden of chronic medical conditions, such as hypertension, heart disease, and diabetes that disproportionately impact individuals living with schizophrenia. Globally, the dramatically reduced life expectancy observed among individuals living with schizophrenia is largely due to preventable and treatable medical conditions. Recent epidemiological studies in India have further observed a mortality rate among individuals living with schizophrenia that is twice the rate observed in the general population, with calls for greater efforts to address this significant health disparity. In addition to recognizing the need to address the alarming care gap, where in India it is estimated that upwards of 75% of individuals living with schizophrenia do not have access to essential mental health care, urgent attention is also needed towards responding to the medical and physical health needs of this vulnerable patient population. Psychosocial interventions, focused on rehabilitation and skill-building, engaging in social activities, managing mental health symptoms, and promoting recovery and community reintegration, hold potential to reduce disability and improve mental health and functioning for individuals living with schizophrenia. Furthermore, building on recent compelling evidence from higher-income countries, community-based programs could be augmented with additional content aimed at addressing risk factors for early mortality, such as lifestyle behaviors, tobacco use, and management of co-occurring chronic medical conditions. Therefore, our study seeks to evaluate the use of a digital platform for supporting the clinical effectiveness and integration of task shared delivery of the evidence-based COPSI (Community care for People with Schizophrenia in India) program in primary care. We will build on important preliminary work led by project collaborators to support our aims to evaluate whether a novel digital platform can enhance the clinical effectiveness (Aim 1) and the integration (Aim 2) of an evidence-based psychosocial rehabilitation intervention for patients with schizophrenia in primary care settings in India.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia per IDC-10 diagnostic criteria for research and an illness duration of greater than 12 months and overall moderate level of severity on the CGI-SCH scale
* At least one risk factor for early mortality (e.g. hypertension, diabetes, dyslipidemia, etc)
* Willingness to stay in the study area during the trial period
* Ability to operate a smartphone

Exclusion Criteria:

* Major visual impairment or inability to operate a smartphone
* Cognitive impairment or diagnosis of dementia
* Planning to move out of the study area in the next 12 months
* Does not speak Hindi or Kannada

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Indian Disability Evaluation and Assessment Scale (IDEAS) | Baseline, 6 months, and 12 months
  - 4-domain self-report measure detecting the level of disability in psychiatric patients in India which generates a global score of severity of disability (0-20) with increasing scores indicating more severe disabilities

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Baseline, 6 months, and 12 months
  30-item self-report measure of positive and negative symptoms and general psychopathology
Generalized Anxiety Disorder Assessment-7 (GAD-7) | Baseline, 6 months, and 12 months
  7-item self-report measure of anxiety symptom severity based on DSM-5 criteria
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 6 months, and 12 months
  9-item self-report measure of depression severity based on DSM-5 criteria
Clinical Global Impression-Schizophrenia (CGI-SCH) Scale | Baseline, 6 months, and 12 months
  7-item self-report measure of severity of schizophrenia, each component of the CGI-SCH is waited separately and does not yield a global score
Brief Assessment of Cognition in Schizophrenia (BACS) | Baseline, 6 months, and 12 months
  Newly developed instrument to assess aspects of cognition in patients with schizophrenia

OTHER OUTCOMES:
Pittsburgh Sleep Questionnaire Index (PSQI) | Baseline, 6 months, and 12 months
  19-item self-report measure of sleep quality for patients with psychiatric disorders
EuroQol-5D (EQ5D) | Baseline, 6 months, and 12 months
  25-item self-report standardized measure of health status and quality of life to provide a generic measure of health for clinical appraisal
Social Functioning Scale (SFS) | Baseline, 6 months, and 12 months
  A measure with 7 subscales used to assess functioning in patients with psychosis
Framingham Risk Score | Baseline, 6 months, and 12 months
  A measure used to assess cardiovascular risk using quantitative information to aid in targeting lower risk factors

CONTACTS AND LOCATIONS:
Overall Officials: John A Naslund, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); John Torous, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Narayana Manjunatha, MD, MBBS, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India

REFERENCES:
- [Background] Tyagi V, Khan A, Siddiqui S, Kakra Abhilashi M, Dhurve P, Tugnawat D, Bhan A, Naslund JA. Development of a Digital Program for Training Community Health Workers in the Detection and Referral of Schizophrenia in Rural India. Psychiatr Q. 2023 Jun;94(2):141-163. doi: 10.1007/s11126-023-10019-w. Epub 2023 Mar 29. PMID 36988785
- [Background] Bondre AP, Shrivastava R, Raghuram H, Tugnawat D, Khan A, Gupta S, Kumar M, Mehta UM, Keshavan M, Lakhtakia T, Chand PK, Thirthalli J, Patel V, Torous J, Rozatkar AR, Naslund JA, Bhan A. A qualitative exploration of perceived needs and barriers of individuals with schizophrenia, caregivers and clinicians in using mental health applications in Madhya Pradesh, India. SSM Ment Health. 2022 Dec;2:100063. doi: 10.1016/j.ssmmh.2022.100063. PMID 36688236
- [Background] Naslund JA, Tyagi V, Khan A, Siddiqui S, Kakra Abhilashi M, Dhurve P, Mehta UM, Rozatkar A, Bhatia U, Vartak A, Torous J, Tugnawat D, Bhan A. Schizophrenia Assessment, Referral and Awareness Training for Health Auxiliaries (SARATHA): Protocol for a Mixed-Methods Pilot Study in Rural India. Int J Environ Res Public Health. 2022 Nov 13;19(22):14936. doi: 10.3390/ijerph192214936. PMID 36429654
- [Background] Lakhtakia T, Bondre A, Chand PK, Chaturvedi N, Choudhary S, Currey D, Dutt S, Khan A, Kumar M, Gupta S, Nagendra S, Reddy PV, Rozatkar A, Scheuer L, Sen Y, Shrivastava R, Singh R, Thirthalli J, Tugnawat DK, Bhan A, Naslund JA, Patel V, Keshavan M, Mehta UM, Torous J. Smartphone digital phenotyping, surveys, and cognitive assessments for global mental health: Initial data and clinical correlations from an international first episode psychosis study. Digit Health. 2022 Nov 8;8:20552076221133758. doi: 10.1177/20552076221133758. eCollection 2022 Jan-Dec. PMID 36386246
- [Background] Rodriguez-Villa E, Rozatkar AR, Kumar M, Patel V, Bondre A, Naik SS, Dutt S, Mehta UM, Nagendra S, Tugnawat D, Shrivastava R, Raghuram H, Khan A, Naslund JA, Gupta S, Bhan A, Thirthall J, Chand PK, Lakhtakia T, Keshavan M, Torous J. Cross cultural and global uses of a digital mental health app: results of focus groups with clinicians, patients and family members in India and the United States. Glob Ment Health (Camb). 2021 Aug 24;8:e30. doi: 10.1017/gmh.2021.28. eCollection 2021. PMID 34512999
- [Background] Rodriguez-Villa E, Mehta UM, Naslund J, Tugnawat D, Gupta S, Thirthalli J, Bhan A, Patel V, Chand PK, Rozatkar A, Keshavan M, Torous J. Smartphone Health Assessment for Relapse Prevention (SHARP): a digital solution toward global mental health - CORRIGENDUM. BJPsych Open. 2021 Feb 5;7(2):e48. doi: 10.1192/bjo.2021.6. No abstract available. PMID 33541463
- [Background] Cohen A, Naslund JA, Chang S, Nagendra S, Bhan A, Rozatkar A, Thirthalli J, Bondre A, Tugnawat D, Reddy PV, Dutt S, Choudhary S, Chand PK, Patel V, Keshavan M, Joshi D, Mehta UM, Torous J. Relapse prediction in schizophrenia with smartphone digital phenotyping during COVID-19: a prospective, three-site, two-country, longitudinal study. Schizophrenia (Heidelb). 2023 Jan 27;9(1):6. doi: 10.1038/s41537-023-00332-5. PMID 36707524